CLINICAL TRIAL: NCT04633447
Title: A Phase 2, Multicenter, Randomized, Placebo-controlled, Double-blind, Proof-of-Concept Study to Evaluate Guselkumab for the Treatment of Participants With New-onset or Relapsing Giant Cell Arteritis
Brief Title: A Study to Evaluate Guselkumab for the Treatment of Participants With New-onset or Relapsing Giant Cell Arteritis
Acronym: THEIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study primary endpoint was not met
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108887; CNTO1959GCA2001 (Other: Janssen Research & Development, LLC); 2020-000622-26 (EudraCT Number)
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Guselkumab (Experimental): Participants will receive guselkumab subcutaneously (SC) every 4 weeks from Week 0 through Wweek 48. This will be in combination with a protocol specified 26-week GC taper. Participants of the long-term extension (LTE) period will continue to receive subcutaneous (SC) injections every 4 weeks starting at Week 52 (LTE Week 0) through Week 100 (LTE Week 48) or until the participants have a Giant cell arteritis (GCA) flare, or the participants discontinues treatment due to unblinding after the Week 60 DBL for the Main study, or until a decision is made not to continue clinical development in this GCA population, whichever occurs first.
  Interventions: Drug: Guselkumab
- Placebo (Experimental): Participants will receive matching placebo SC every 4 weeks from Week 0 through Week 48. This will be in combination with a protocol-specified 26-week GC taper. Participants of the LTE period will continue to receive SC injections every 4 weeks starting at Week 52 (LTE Week 0) through Week 100 (LTE Week 48) or until the participants have a GCA flare, or the participants discontinues treatment due to unblinding after the Week 60 DBL for the Main study, or until a decision is made not to continue clinical development in this GCA population, whichever occurs first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered subcutaneously.
  Other Names: Tremfya; CNTO 1959
  Arms: Guselkumab
Drug: Placebo — Matching placebo will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of guselkumab compared to placebo, in combination with a 26-week glucocorticoid (GC) taper regimen, in adult participants with new-onset or relapsing giant cell arteritis (GCA).

DETAILED DESCRIPTION:
Giant cell arteritis (GCA) is a non-necrotizing granulomatous systemic vasculitis of unknown etiology affecting medium-sized and large arteries usually accompanied or preceded by systemic inflammation. Guselkumab is a monoclonal antibody (mAb) that binds to the p19 sub-unit of human interleukin (IL)-23 with high affinity and blocks binding of extracellular IL-23 to cell surface IL-23 receptor, inhibiting IL 23 specific intracellular signaling and subsequent activation and cytokine production. It is used in treatment of psoriatic arthritis, generalized pustular psoriasis, erythrodermic psoriasis. The study consists of a screening period (less than or equal to [<=] 6 weeks), double-blind treatment period (48 weeks), and safety follow-up period (12 weeks). Participants who complete the Week 52 visit and are assessed to be in glucocorticoid (GC)-free remission, may have the option to participate in the long-term extension (LTE) period of the study for up to 12 months. This study will evaluate the efficacy, safety, Pharmacokinetics (PK), and immunogenicity of guselkumab in combination with a 26-week GC taper regimen for the treatment of active new-onset or relapsing GCA in adult participants. The total duration of the study is up to 66 weeks for the main study and for participants that continue in the LTE period, the total study duration will be up to 112 weeks.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of Giant cell arteritis (GCA) according to the revised American College of Rheumatology criteria
* GCA diagnosis confirmed by either temporal artery biopsy revealing features of GCA either at time of diagnosis or at other timepoint during disease history; or evidence of cranial GCA either at time of diagnosis or at other timepoint during disease history by cranial doppler-ultrasound; or cranial Magnetic Resonance Imaging (MRI) or Magnetic Resonance Angiography; or other imaging modality upon agreement with the sponsor or evidence of GCA by angiography or cross-sectional imaging (ultrasound, MRI, computed tomography [CT], positron emission tomography [PET])
* Have new onset or relapsing GCA
* Have active GCA within 6 weeks of first study intervention: Active GCA: presence of signs and symptoms of GCA and elevated erythrocyte sedimentation rate (ESR) greater than or equal to (>=) 30 millimeter per hour (mm/hour), or C-reactive protein (CRP) >= 10 milligrams per liter (mg/L) (or 1 milligrams per deciliter [mg/dL]), attributed to active GCA. ESR >= 30 mm/hour or CRP >= 10 mg/L (or 1 mg/dL) is not required if active GCA has been confirmed by a positive temporal artery biopsy or ultrasound or other imaging modality within 6 weeks of first study intervention
* Clinically stable GCA disease on a glucocorticoid (GC) dose between 20 and 60 milligrams per day (mg/day) (prednisone or equivalent) at randomization such that the participant is able to safely participate in the protocol defined prednisone taper regimen, in the opinion of the investigator

Exclusion criteria

* Has any known severe or uncontrolled GCA complications
* Has any rheumatic disease other than GCA such that could interfere with assessment of GCA
* Has a current diagnosis or signs or symptoms of severe, progressive, or concomitant medical condition that places the participant at risk by participating in this study)
* Has or has had any major ischemic event, within 12 weeks of first study intervention. Has a personal history of arterial thrombosis or venous thromboembolism (including deep venous thrombosis [DVT] and Pulmonary Embolism [PE])
* Has any comorbidities requiring 3 or more courses of systemic GCs within 12 months of first study intervention, AND, inability, in the opinion of the investigator, to withdraw GC therapy through protocol-defined taper regimen due to suspected or established adrenal insufficiency, OR, currently on systemic chronic GC therapy for reasons other than GCA and be GC dependent and have the potential to flare due to GC tapering (e.g. unstable asthma, unstable COPD)
* Has a history of, or ongoing, chronic or recurrent infectious disease
* Has received within specified timeframe, or 5 half-lives (whichever is greater) , or has failed treatment with any investigational or approved biologic agents or Janus Kinase Inhibitor prior to first study intervention
* Use of any of the following systemic immunosuppressant treatments within the specified timeframe prior to study start: Any cytotoxic agents (cyclophosphamide, chlorambucil, nitrogen mustard, or other alkylating agents) with 6 months; Hydroxychloroquine, cyclosporine A, azathioprine, tacrolimus, sirolimus, sulfasalazine, leflunomide with cholestyramine washout or mycophenolate mofetil/mycophenolic acid within 3 months; Intramuscular, intra-articular, intrabursal, epidural, intra-lesional or IV GCs within 6 week; and Methotrexate (MTX) within 12 weeks. If started MTX >12 weeks prior to first study intervention MTX must have been at a stable dose for minimally 4 weeks and must not be receiving more than 25 mg oral or SC MTX per week
* Has chronic continuous use of systemic GCs for greater than (>) 4 years or inability, in the opinion of the investigator, to withdraw GC treatment through protocol-defined taper regimen due to suspected or established adrenal insufficiency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (30):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- France (2):
  - CHU Dijon, Dijon
  - Hopital Cochin, Paris
- Germany (3):
  - Universitatsklinikum Erlangen, Erlangen
  - medius KLINIK KIRCHHEIM, Kirchheim unter Teck
  - Universitatsklinik Tubingen, Tübingen
- Israel (4):
  - Bnai Zion Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Azianeda Ospedaliera dell'alto adige - Ospedale di Brunico, Bolzano
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda USL 4 Prato, Prato
  - ASUI Santa Maria della Misericordia di Udine, Udine
- Poland (3):
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
  - Szpital Specjalistyczny im. J. Dietla, Krakow
  - NZOZ Lecznica MAK MED S C, Nadarzyn
- Spain (6):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. Marques de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Guselkumab: Initially, subjects received 3 intravenous (IV) induction doses of Guselkumab 400 milligrams (mg) every 4 weeks starting from Week 0 up to Week 8 followed by a subcutaneous (SC) maintenance regimen of Guselkumab 200 mg every 4 weeks starting from Week 12 until Week 48 in the main study along with a protocol defined 26-week Glucocorticoid (GC) taper regimen. Subjects were then followed up for safety for 12 weeks until Week 60. With protocol amendment 5, IV induction was discontinued, and subjects enrolled from that point onwards received Guselkumab 200 mg subcutaneously every 4 weeks Week 0 until Week 48 (end of treatment). Eligible subjects who were in GC-free remission at Week 48 and consented for the long term extension (LTE) period, continued to receive Guselkumab 200 mg subcutaneously every 4 weeks starting from Week 52 (LTE Week 0) until Week 100 (LTE Week 48). Subjects were then followed up for safety for 12 weeks after the last dose up to Week 112. Participants who did not enter LTE continued in the main study till Week 60.
- Placebo: Initially, participants received 3 IV induction doses of Placebo matching to Guselkumab 400 mg every 4 weeks starting from Week 0 up to Week 8 followed by a SC maintenance regimen of placebo matching to Guselkumab 200 mg every 4 weeks starting from Week 12 until Week 48 in the main study along with a protocol defined 26-week GC taper regimen. Participants were then followed up for safety for 12 weeks until Week 60. With protocol amendment 5, IV induction was discontinued, and participants enrolled from that point onwards received placebo matching to guselkumab 200 mg subcutaneously every 4 weeks from Week 0 until Week 48 (end of treatment). Eligible participants who were in GC-free remission at Week 48 and consented for the LTE period, continued to receive placebo matching to guselkumab 200 mg subcutaneously every 4 weeks starting from Week 52 (LTE Week 0) until Week 100 (LTE Week 48). Participants were then followed up for safety for 12 weeks after the last dose up to Week 112. Participants who did not enter LTE continued in the main study till Week 60.
Period: Main Study (From Week 0 up to Week 60)
Arm/Group | Guselkumab | Placebo
Started | 35 | 18
Participants Enrolled Post PA-5 Who Received Placebo Matching to Guselkumab 200 mg From Week 0 | 0 | 11
Participants Enrolled Post PA-5 Who Received Guselkumab 200 mg From Week 0 | 19 | 0
Completed | 22 | 12
Not Completed | 13 | 6
Not completed — Adverse Event | 8 | 2
Not completed — Study terminated by sponsor | 3 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Period: LTE Period (Week 52 up to Week 112)
Arm/Group | Guselkumab | Placebo
Started | 9 | 6
Completed | 5 | 3
Not Completed | 4 | 3
Not completed — Study Terminated by Sponsor | 3 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guselkumab | Placebo | Total
Number analyzed (Participants) | 35 | 18 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 29 | 15 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (7.65) | 70.8 (7.14) | 71.5 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 37
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 27 | 15 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 18 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4 | 0 | 4
  Canada | 8 | 4 | 12
  France | 3 | 0 | 3
  Germany | 2 | 3 | 5
  Israel | 3 | 1 | 4
  Italy | 5 | 5 | 10
  Poland | 2 | 0 | 2
  Spain | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Percentage of Participants Achieving Glucocorticoid (GC)-Free Remission at Week 28
Description: GC free remission at Week 28 was defined as (1) no signs or symptoms of active Giant cell arteritis (GCA) at Week 28; (2) absence of GCA flare from first dose of the study drug through Week 28; and (3) adherence to the protocol specified 26-week GC taper regimen. GCA flare was defined as the recurrence of signs and symptoms of active GCA, with or without elevation of inflammatory markers, and with the necessity for an increase in GC dose for GCA.
Time Frame: Week 28
Population: Full analysis set (FAS) included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of Participants
Groups:
- Main Study: Guselkumab: Initially, participants received 3 intravenous (IV) induction doses of Guselkumab 400 milligrams (mg) every 4 weeks starting from Week 0 up to Week 8 followed by a subcutaneous (SC) maintenance regimen of Guselkumab 200 mg every 4 weeks starting from Week 12 until Week 48 in the main study along with a protocol defined 26-week Glucocorticoid (GC) taper regimen. Participants were then followed up for safety for 12 weeks until Week 60. With protocol amendment 5, IV induction was discontinued, and participants enrolled from that point onwards received Guselkumab 200 mg subcutaneously every 4 weeks from Week 0 until Week 48 (end of treatment). Participants who did not enter LTE continued in the main study till Week 60.
- Main Study: Placebo: Initially, participants received 3 IV induction doses of Placebo matching to Guselkumab 400 mg every 4 weeks starting from Week 0 up to Week 8 followed by a SC maintenance regimen of placebo matching to Guselkumab 200 mg every 4 weeks starting from Week 12 until Week 48 in the main study along with a protocol defined 26-week GC taper regimen. Participants were then followed up for safety for 12 weeks until Week 60. With protocol amendment 5, IV induction was discontinued, and participants enrolled from that point onwards received placebo matching to guselkumab 200 mg subcutaneously every 4 weeks from Week 0 until Week 48 (end of treatment). Participants who did not enter LTE continued in the main study till Week 60.
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Percentage of Participants | 40.0 | 33.3
Statistical Analysis 1: Comparison: Main Study: Guselkumab vs Main Study: Placebo; Test type: Superiority; p = 0.638, Cochran-Mantel-Haenszel; Difference in Percentage = 6.6, 90% CI 2-sided [-14.7 to 27.9]

2. Secondary Outcome: Main Study: Percentage of Participants Achieving GC-Free Remission at Weeks 28, 32, 36, 40, 44, 48 and 52
Description: GC free remission was defined as (1) no signs or symptoms of active GCA at Weeks 28, 32, 36, 40, 44, 48 and 52 respectively; (2) absence of GCA flare from first dose of the study drug through Weeks 28, 32, 36, 40, 44, 48 and 52; (3) adherence to the protocol specified 26-week GC taper regimen. GCA flare was defined as the recurrence of signs and symptoms of active GCA, with or without elevation of inflammatory markers, and with the necessity for an increase in GC dose for GCA.
Time Frame: Weeks 28, 32, 36, 40, 44, 48 and 52
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Percentage of Participants
  At Week 28 | 40.0 | 33.3
  At Week 32 | 34.3 | 33.3
  At Week 36 | 34.3 | 33.3
  At Week 40 | 34.3 | 33.3
  At Week 44 | 34.3 | 33.3
  At Week 48 | 31.4 | 27.8
  At Week 52 | 25.7 | 27.8

3. Secondary Outcome: Main Study: Percentage of Participants Achieving Both GC-Free Remission and Normalization of Erythrocyte Sedimentation Rate (ESR) at Weeks 28, 32, 36, 40, 44, 48 and 52
Description: GC-free remission at Weeks 28, 32, 36, 40, 44, 48 and 52 was defined as (1) no signs or symptoms of active GCA at Weeks 28, 32, 36, 40, 44, 48 and 52 respectively (2) absence of GCA flare from first dose of the study drug through Weeks 28, 32, 36, 40, 44, 48 and 52 (3) adherence to the protocol specified 26-week GC taper regimen. Normalization of ESR was defined as ESR less than (<) 30 millimeter per hour (mm/hr) at Weeks 28, 32, 36, 40, 44, 48 and 52. GCA flare was defined as the recurrence of signs and symptoms of active GCA, with or without elevation of inflammatory markers, and with the necessity for an increase in GC dose for GCA.
Time Frame: Weeks 28, 32, 36, 40, 44, 48 and 52
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Percentage of Participants
  At Week 28 | 22.9 | 5.6
  At Week 32 | 22.9 | 11.1
  At Week 36 | 22.9 | 16.7
  At Week 40 | 25.7 | 16.7
  At Week 44 | 22.9 | 11.1
  At Week 48 | 20.0 | 22.2
  At Week 52 | 22.9 | 16.7

4. Secondary Outcome: Main Study: Percentage of Participants Achieving Both GC-Free Remission and Normalization of C-Reactive Protein (CRP) at Weeks 28, 32, 36, 40, 44, 48 and 52
Description: GC-free remission at Weeks 28, 32, 36, 40, 44, 48 and 52 was defined as (1) no signs or symptoms of active Giant cell arteritis (GCA) at Weeks 28, 32, 36, 40, 44, 48 and 52 respectively (2) absence of GCA flare from first dose of the study drug through Weeks 28, 32, 36, 40, 44, 48 and 52 (3) adherence to the protocol specified 26-week GC taper regimen. Normalization of CRP is defined as CRP <10 milligrams per liter (mg/L) or <1 milligrams per deciliter (mg/dL). GCA flare was defined as the recurrence of signs and symptoms of active GCA, with or without elevation of inflammatory markers, and with the necessity for an increase in GC dose for GCA.
Time Frame: Weeks 28, 32, 36, 40, 44, 48 and 52
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Percentage of Participants
  At Week 28 | 22.9 | 16.7
  At Week 32 | 20.0 | 16.7
  At Week 36 | 25.7 | 22.2
  At Week 40 | 28.6 | 33.3
  At Week 44 | 25.7 | 27.8
  At Week 48 | 20.0 | 27.8
  At Week 52 | 17.1 | 22.2

5. Secondary Outcome: Main Study: Percentage of Participants Achieving Both GC-Free Remission and Normalization of Both ESR and CRP at Weeks 28, 32, 36, 40, 44, 48 and 52
Description: GC-free remission at Weeks 28, 32, 36, 40, 44, 48 and 52 was defined as (1) no signs or symptoms of active GCA at Weeks 28, 32, 36, 40, 44, 48 and 52 respectively; (2) absence of GCA flare from first dose of the study drug through Weeks 28, 32, 36, 40, 44, 48 and 52; (3) adherence to the protocol specified 26-week GC taper regimen. Normalization of ESR is defined as ESR < 30 mm/hr at Weeks 28, 32, 36, 40, 44, 48 and 52. Normalization of CRP is defined as CRP <10 mg/L or <1 mg/dL. GCA flare was defined as the recurrence of signs and symptoms of active GCA, with or without elevation of inflammatory markers, and with the necessity for an increase in GC dose for GCA.
Time Frame: Weeks 28, 32, 36, 40, 44, 48 and 52
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Percentage of Participants
  At Week 28 | 14.3 | 5.6
  At Week 32 | 17.1 | 11.1
  At Week 36 | 20.0 | 16.7
  At Week 40 | 22.9 | 16.7
  At Week 44 | 17.1 | 11.1
  At Week 48 | 14.3 | 22.2
  At Week 52 | 17.1 | 16.7

6. Secondary Outcome: Main Study: Cumulative Glucocorticoid (GC) Dose
Description: Total cumulative GC dose administered included GCA taper, GC rescue therapy as well as for all other indications (any oral GC) from baseline (Day 1) up to Weeks 28 and 52 was reported.
Time Frame: Baseline (Day 1) up to Weeks 28 and 52
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Median (Full Range); unit: Milligrams (mg)
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Milligrams (mg)
  Baseline (Day 1) up to Week 28 | 2231.0 [1315 to 4146] | 2205.0 [1736 to 6010]
  Baseline (Day 1) up to Week 52 | 2418.5 [1315 to 4319] | 2902.1 [1736 to 7345]

7. Secondary Outcome: Main Study: Time to First GCA Disease Flare or Discontinuation of Study Intervention Due to Adverse Event (AE) of Worsening of GCA
Description: Time to occurrence of GCA disease flare was defined as the time from first dose of the study agent to the occurrence of the first observation of GCA disease flare or discontinuation due to adverse event (AE) of worsening of GCA. GCA flare was defined as the recurrence of signs and symptoms of active GCA, with or without elevation of inflammatory markers, and with the necessity for an increase in GC dose for GCA.
Time Frame: Baseline (Day 1) up to Week 30 and Week 52
Population: FAS included all randomized participants who received at least 1 administration of study intervention. Here, N (Overall Number of Participants analyzed) signifies participants with at least 1 disease flare or discontinuation of study intervention due to AE of Worsening of GCA.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Weeks
  Baseline (Day 1) up to Week 30 | NA [27.71 to NA] — Median and upper limit of 90% confidence interval (CI) could not be estimated due to low number of participants with events. | 29.71 [20.14 to NA] — Upper limit of 90% CI could not be estimated due to low number of participants with events.
  Baseline (Day 1) up to Week 52 | NA [27.71 to NA] — Median and upper limit of 90% CI could not be estimated due to low number of participants with events. | 30.07 [20.14 to NA] — Upper limit of 90% CI could not be estimated due to low number of participants with events.

8. Secondary Outcome: Main Study: Number of Participants With GCA Disease Flares or Discontinuation of Study Intervention Due to AE of Worsening of GCA
Description: Number of participants with GCA disease flares or discontinuation of study intervention due to AE of worsening of GCA were reported. GCA flare was defined as the recurrence of signs and symptoms of active GCA, with or without elevation of inflammatory markers, and with the necessity for an increase in GC dose for GCA.
Time Frame: Baseline (Day 1) up to Week 30 and Week 52
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Participants
  Baseline up to Week 30: 1 Flare | 10 | 8
  Baseline up to Week 30: 2 Flares | 0 | 0
  Baseline up to Week 30: >=3 Flares | 0 | 0
  Baseline up to Week 52: 1 Flare | 13 | 7
  Baseline up to Week 52: 2 Flares | 3 | 3
  Baseline up to Week 52: >=3 Flares | 0 | 0

9. Secondary Outcome: Main Study: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs (including serious and non-serious AEs) were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Any AE occurring at or after the initial administration of study intervention through the end of the main study was considered to be treatment emergent.
Time Frame: Baseline (Day 1) up to Week 60
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Participants | 34 | 17

10. Secondary Outcome: Number of Participants With TEAEs by System Organ Class (SOC) With a Frequency Threshold of 5 Percent (%) or More
Description: Number of participants with TEAEs (including serious and non-serious AEs) by SOC with a frequency threshold of 5 percent (%) or more were reported. An adverse event (AE) was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Any AE occurring at or after the initial administration of study intervention through the end of the main study was considered to be treatment emergent.
Time Frame: Baseline (Day 1) up to Week 60
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Participants
  Infections and infestations | 21 | 11
  Musculoskeletal and connective tissue disorders | 19 | 5
  Vascular disorders | 18 | 11
  Gastrointestinal disorders | 10 | 2
  General disorders and administration site conditions | 10 | 6
  Nervous system disorders | 9 | 9
  Eye disorders | 8 | 3
  Respiratory, thoracic and mediastinal disorders | 8 | 4
  Skin and subcutaneous tissue disorders | 8 | 1
  Injury, poisoning and procedural complications | 7 | 2
  Investigations | 6 | 0
  Endocrine disorders | 5 | 0
  Psychiatric disorders | 4 | 1
  Metabolism and nutrition disorders | 3 | 1
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 3 | 1
  Cardiac disorders | 2 | 2
  Renal and urinary disorders | 2 | 1
  Reproductive system and breast disorders | 1 | 1

11. Secondary Outcome: Main Study: Number of Participants With Treatment-emergent Serious Adverse Event (SAEs)
Description: Number of participants with treatment emergent SAEs were reported. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurred at or after the initial administration of study intervention through the end of the main study was considered to be treatment emergent.
Time Frame: Baseline (Day 1) up to Week 60
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Participants | 6 | 0

12. Secondary Outcome: Main Study: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Number of participants with clinically significant abnormalities in vital signs were reported. Clinically significant abnormal vital signs criteria: Pulse rate: <50 beats per minutes (bpm) and with greater than (>) 20 bpm decrease from baseline, >115 bpm and with >30 bpm increase from baseline; Systolic blood pressure (SBP): <90 millimeters of mercury [mmHg] and with >30 mmHg decrease from baseline, >150 mmHg and with >40 mmHg increase from baseline; Diastolic blood pressure (DBP): <50 mmHg and with >20 mmHg decrease from baseline, >95 mmHg and with >30 mmHg increase from baseline; Interarm blood pressure: Interarm blood pressure difference greater than or equal to (>=) 15 mmHg in systolic blood pressure at 3 consecutive visits; Temperature (Temp): >38.4 Degree Celsius (C) and with >=1 C increase from baseline; Weight (kilogram [kg]): decrease 10 percent (%) from baseline, increase 10% from baseline; Respiratory Rate: >20 breaths per minute.
Time Frame: Baseline (Day 1) up to Week 60
Population: Safety analysis set included all participants who received at least 1 dose of study intervention and had at least one post baseline value for the specified vital sign parameter. Here, "n"(number analyzed) signifies number of participants analyzed at specified categories
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Participants
  Pulse rate: <50 bpm and with >20 bpm decrease | 1 | 0
  Pulse rate: >115 bpm and with >30 bpm increase | 0 | 0
  Systolic BP: <90 mmHg and >30 mmHg decrease | 2 | 0
  Systolic BP: >150 mmHg and >40 mmHg increase | 0 | 2
  Diastolic BP: <50 mmHg and >20 mmHg decrease | 2 | 0
  Diastolic BP: >95 mmHg and >30 mmHg increase | 1 | 1
  Interarm BP:BP difference >=15 mmHg in systolic BP | 2 | 2
  Temp: >38.4 C and >=1 C increase from baseline | 0 | 0
  Weight: Decrease 10% from baseline: number analyzed (Participants) | 30 | 18
  Weight: Decrease 10% from baseline | 0 | 1
  Weight: Increase 10% from baseline: number analyzed (Participants) | 30 | 18
  Weight: Increase 10% from baseline | 6 | 2
  Respiratory Rate: >20 breaths per minute | 1 | 4

13. Secondary Outcome: Main Study: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Number of participants with National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade 3 or 4 abnormalities in clinical laboratory tests: hematology and chemistry were reported. Clinical laboratory abnormalities of living participants were assessed as per NCI CTCAE version 5, grades (0-4), where Grade 0-Normal, Grade 1- Mild, Grade 2- Moderate, Grade 3- Severe or medically significant but not immediately life-threatening, Grade 4- Life-threatening consequences. Higher grades showed severe abnormality. As per the discretion of investigator, laboratory abnormalities with NCI CTCAE Grade 3 or 4 were considered clinically significant. Combined data of Grade 3 and 4 abnormalities are reported as planned. Only those categories in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to Week 60
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Guselkumab | Main Study: Placebo
Number analyzed (Participants) | 35 | 18
Participants
  Chemistry: Creatinine Increased | 1 | 0
  Chemistry: Alanine Aminotransferase Increased | 1 | 0
  Hematology: Lymphocyte Count Decreased | 3 | 3

14. Secondary Outcome: Main Study: Serum Concentrations of Guselkumab
Description: Serum concentrations of Guselkumab over time was reported.
Time Frame: Pre-dose and 1 hour post dose on Week 0 (Day 1), Week 4 (Day 28), and Week 8 (Day 56); Week 12 (Day 84), Week 16 (Day 112), Week 28 (Day 196), Week 52 (Day 364)
Population: Pharmacokinetics (PK) analysis set included all participants who received at least 1 administration of Guselkumab and had at least one valid post dose blood sample drawn for PK analysis. Here, N (Overall number of participant analyzed) signifies number of participant evaluable for this outcome measure and n (number analyzed) signifies number of participants evaluable at specified timepoints. This outcome measure was planned to be analyzed for Guselkumab arm only.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL
Arm/Group | Main Study: Guselkumab
Number analyzed (Participants) | 35
Microgram per milliliter (mcg/mL
  Pre dose on Week 0 (Day 1): number analyzed (Participants) | 34
  Pre dose on Week 0 (Day 1) | 0.00 (0.000)
  1 Hour Post Dose on Week 0 (Day 1): number analyzed (Participants) | 15
  1 Hour Post Dose on Week 0 (Day 1) | 130.93 (45.522)
  Pre dose on Week 4 (Day 28): number analyzed (Participants) | 32
  Pre dose on Week 4 (Day 28) | 11.21 (6.616)
  1 Hour Post Dose on Week 4 (Day 28): number analyzed (Participants) | 12
  1 Hour Post Dose on Week 4 (Day 28) | 150.21 (34.952)
  Pre dose on Week 8 (Day 56): number analyzed (Participants) | 30
  Pre dose on Week 8 (Day 56) | 19.71 (23.002)
  1 Hour Post Dose on Week 8 (Day 56): number analyzed (Participants) | 9
  1 Hour Post Dose on Week 8 (Day 56) | 127.14 (68.157)
  Week 12 (Day 84): number analyzed (Participants) | 31
  Week 12 (Day 84) | 19.16 (17.831)
  Week 16 (Day 112): number analyzed (Participants) | 29
  Week 16 (Day 112) | 15.81 (9.644)
  Week 28 (Day 196): number analyzed (Participants) | 25
  Week 28 (Day 196) | 12.63 (4.824)
  Week 52 (Day 364): number analyzed (Participants) | 19
  Week 52 (Day 364) | 12.55 (4.701)

15. Secondary Outcome: Main Study: Number of Participants With Antibodies to Guselkumab
Description: Number of participants with antibodies to Guselkumab were reported.
Time Frame: Baseline (Day 1) up to Week 28, Week 52
Population: Immunogenicity analysis set included all participants who received at least 1 administration of guselkumab and have at least one post-dose sample collection. This outcome measure was planned to be analyzed for Guselkumab arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Guselkumab
Number analyzed (Participants) | 35
Participants
  Baseline (Day 1) up to Week 28 | 1
  Baseline (Day 1) up to Week 52 | 3

ADVERSE EVENTS:
Time Frame: Main study: All-Cause Mortality: From Screening (-6 weeks) up to Week 60; SAEs & Other AEs: Baseline (Day 1) up to Week 60. LTE Period: From Week 52 (LTE Week 0) up to Week 112 (LTE Week 60)
Description: Safety analysis set included all subjects who received at least 1 dose of study intervention.
Groups:
- LTE Period: Guselkumab: At Week 48, participants from main study who were in GC-free remission and consented for the long term extension (LTE) period, continued to receive Guselkumab 200 mg subcutaneously every 4 weeks starting from Week 52 (LTE Week 0) until Week 100 (LTE Week 48). Participants were then followed up for safety for 12 weeks after the last dose up to Week 112.
- LTE Period: Placebo: At Week 48, participants from main study who were in GC-free remission and consented for the LTE period, continued to receive placebo matching to guselkumab 200 mg subcutaneously every 4 weeks starting from Week 52 (LTE Week 0) until Week 100 (LTE Week 48). Participants were then followed up for safety for 12 weeks after the last dose up to Week 112.
Arm/Group | Main Study: Guselkumab | Main Study: Placebo | LTE Period: Guselkumab | LTE Period: Placebo
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/18 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/35 | 0/18 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 31/35 | 17/18 | 6/9 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Guselkumab (N=35) | Main Study: Placebo (N=18) | LTE Period: Guselkumab (N=9) | LTE Period: Placebo (N=6)
Abdominal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Peripheral Artery Stenosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Guselkumab (N=35) | Main Study: Placebo (N=18) | LTE Period: Guselkumab (N=9) | LTE Period: Placebo (N=6)
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 2 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 2 | 1 | 0 | 0
Cataract Nuclear (Eye disorders) | 0 | 1 | 0 | 0
Macular Degeneration (Eye disorders) | 0 | 0 | 1 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0
Visual Field Defect (Eye disorders) | 2 | 0 | 0 | 0
Abdominal Mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 0 | 0
Complication Associated with Device (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 2 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 1 | 0 | 0
Peripheral Swelling (General disorders) | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 1 | 0
Covid-19 (Infections and infestations) | 8 | 5 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 2 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 1 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 4 | 2 | 0 | 0
Tinea Pedis (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 2 | 0 | 0 | 0
Weight Increased (Investigations) | 2 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Greater Trochanteric Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain Fog (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness Postural (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 7 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Haemorrhage Urinary Tract (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Skin Fragility (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0
Giant Cell Arteritis (Vascular disorders) | 17 | 10 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04633447/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04633447/SAP_001.pdf